CLINICAL TRIAL: NCT06905405
Title: Assessing the Ability to Improve the Diagnosis of Heart Failure With Preserved Ejection Fraction Using Advanced Imaging Techniques
Brief Title: The Use of Advanced Imaging in HFpEF
Status: Not yet recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH 23163; 232436D (Other Grant/Funding Number: Sheffield Hospitals Charity)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No therapy intervention: cMRI & TTE, no further intervention
  Interventions: Diagnostic Test: Advanced imaging
- Therapy intervention: cMRI & TTE, SGLT-2 inhibitor therapy
  Interventions: Diagnostic Test: Advanced imaging; Drug: SGLT-2 inhibitor

INTERVENTIONS:
Diagnostic Test: Advanced imaging — Cardiac MRI scan Transthoracic ECHO
  Other Names: TTE; cMRI
Drug: SGLT-2 inhibitor — SGLT-2 inhibitor
  Groups: Therapy intervention

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) causes symptoms of breathlessness and leg swelling. It is associated with significant number of hospital admissions and could lead to the patient's death. In HFpEF, the pumping function of the heart is normal but the heart is too stiff to fill properly. The first line investigation is an ultrasound of the heart (echocardiography). A number of parameters are assessed that indicate stiffness within the heart or raised pressures within the heart. However, most of these parameters lack sensitivity which can make HFpEF difficult to diagnose. The best test is to invasively measure the pressures in the heart at rest and with exercise in a procedure called heart catheterisation. However, this is invasive and not readily available. As a result, HFpEF is significantly under diagnosed meaning many patients do not get access to disease specific treatment that may improve symptoms and quality of life. There are a number of new imaging techniques that may help us to better identify HFpEF . However, it is not currently known how to best apply them in clinical practice.

In this study, the investigators will recruit patients presenting to the HF clinic at Sheffield Teaching Hospitals who have symptoms of HFpEF but whose diagnosis remains unclear after initial assessment. The impact of their symptoms will be assessed with the use of a quality of life (QoL) questionnaires and a six-minute walk test (6MWT). They will undergo advanced imaging with a specialist echocardiogram and a cardiac MRI scan. If they are found to have features of HFpEF, they will be started on disease specific treatment. All patients will be followed up after six months to see if they have any symptomatic or functional improvement. They will also undergo repeat imaging to see if there has been any change in the imaging parameters.

DETAILED DESCRIPTION:
The investigators will recruit patients from the Diagnostic heart failure (HF) clinic at Northern General Hospital, Sheffield. Patients with symptoms suggestive of HF but with an indeterminate diagnosis after standard assessment will be recruited.

They will be assessed against the following inclusion and exclusion criteria. Inclusion criteria: Male or female > 18yrs of age. Symptoms of shortness of breath on exertion. NTproBNP (blood test of heart failure) >400 ng/L in sinus rhythm (SR). Baseline TTE demonstrating a dilated left atrium (LA>34 ml/m2), but that otherwise does not meet the current criteria for the diagnosis of HF.

Exclusion criteria: Inability to give informed consent. History of HF, contraindications to SGLT2 inhibitor (a history of type 1 diabetes mellitus, ketoacidosis, allergy to SGLT2 inhibitors, planned or current use of SGLT2 inhibitors or active genital infection). Atrial Fibrillation. Current history of anginal chest pain. All patients will provide written informed consent.

Upon recruitment, all patients will be invited to complete a quality of life questionnaire to assess the burden of their symptoms. The EQ-5Q-5L and KCCQ questionnaires will be used which have widely been used in this patient group.

At the same visit, patients will also undergo a 6-minute walk test (6MWT), repeated twice to mitigate the 'training' effect.

This will document the exercise capacity of the patient in a standard, reproducible, and universally achievable way.

All patients will have already undergone standard echocardiographic imaging as part of their clinical diagnostic work up (cardiac ultrasound). These images will be reviewed by RG (PI) to determine their suitability for advanced analysis.

In this study, the investigators want to assess a novel parameter called atrial strain. This can be performed offline after the procedure but requires good quality images. In many cases, this will be possible without the patient having to undergo further imaging. However, the investigators predict that approximately 25% of cases will require additional images to be obtained.

Where this in the case, patients will be invited back for a further, targeted cardiac ultrasound scan that will be performed by the PI. The investigators will endeavour to perform this at the same visit as the 6MWT to reduce the number of appointments.

Following this, all participants will undergo a cardiac magnetic resonance imaging (MRI) scan on the University of Sheffield CMR scanner. This will include the administration of contrast and a stress drug (regadenason). The purpose of this is to examine the blood supply to the heart as well as the heart function. The whole scan will take approximately one hour. Multiple parameters will be assessed which are detailed in the study protocol.

Once patients have undergone both imaging studies (cardiac ultrasound and cardiac MRI), the results will be reviewed together by the co-investigators (RG and AAM). RG is an experienced cardiac ultrasound and cardiac MRI reporter and AAM is an experienced HF and imaging consultant. The imaging diagnosis of HFpEF is complex and there are a large number of parameters being assessed. As such, results from both the tests with be considered together and consensus researched between the Co-Is as to the likelihood of a diagnosis of HF. The investigators estimate that 25% of participants will have features of HF on these advanced imaging techniques.

Patients with features of HF identified will be commenced on disease specific treatment (SGLT2i therapy) in keeping with current guidelines for the treatment of HF. Patients will receive appropriate counselling and monitoring in keeping with standard clinical practice. Patients without features of HF will not be started on SGLT2i therapy and any further investigation or management will be guided by their clinical history in keeping with standard clinical practice.

Follow up visit (approximately 6 months) All patients will be followed up at 6 months from their initial baseline visit. At this visit they will undergo repeat 6MWT, QoL questionnaires and reassessment of NT pro BNP levels (blood test marker of HF). Patients that were started on disease specific treatment will also undergo repeat imaging. The CMR will not be repeated if no abnormalities were found on the baseline scan. Where the CMR is to be repeated this will can done on the same day or arranged for a different day depending on patient preference. Patients that did not have features of HFpEF and therefore were not started on treatment will not undergo any further imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18yrs of age.
* Symptoms of dysponea on exertion.
* NTproBNP >400 ng/L in sinus rhythm (SR).
* Baseline TTE demonstrating a dilated LA (LA>34 ml/m2), but that otherwise does not meet the current criteria for the diagnosis of HFpEF or HFrEF (preserved LV systolic function, Normal E/e', no evidence of LVH, Estimated PAP < 35mmhg).

Exclusion Criteria:

* Inability to give informed consent. History of HFrEF
* contraindications to SGLT2 inhibitor (a history of type 1 diabetes mellitus, ketoacidosis, allergy to SGLT2 inhibitors, planned or current use of SGLT2 inhibitors or active genital infection).
* Atrial Fibrillation.
* Current history of anginal chest pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to a cardiology clinic with symptoms that may be suggestive of HFpEF, such as breathlessness or fluid overload, but who didn't meet the criteria for diagnosis based on standard imaging.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 18 months
  The number (proportion) of patients presenting to the HF clinic who do not currently meet the standard criteria for the diagnosis of HFpEF based on standard TTE assessment that have evidence of HFpEF on advanced imaging.

SECONDARY OUTCOMES:
Secondary Outcome | 18 months
  As a secondary outcome, we will assess the relationship (correlation) between advanced imaging metrics and QoL and exercise capacity. The following metrics will be assessed:
  * Imaging outcome measures (TTE derived, CMR derived)
  * Clinical outcome measures (6MWT / KCCQ QoL / EQ-5D-5L QoL)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sheffield, Sheffield, United Kingdom